CLINICAL TRIAL: NCT03403283
Title: Dyslipidemia and Diabetic Retinopathy
Acronym: D&D
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Maria Grant, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: 300000188; 5R01EY016077 (NIH)
Record Dates: First submitted 2014-08-07; First posted 2018-01-18 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Retinopathy; Dyslipidemia
MeSH Terms: conditions — Diabetic Retinopathy; Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetic: Diabetics with mild, moderate or severe non proliferative retinopathy and proliferative retinopathy
  Interventions: Other: 15 subjects with Non Proliferative Diabetic Retinopathy(mild, moderate and severe). 15 subjects with Proliferative Diabetic Retinopathy
- Controls: Healthy Controls
  Interventions: Other: Healthy Controls 15 age matched control subjects

INTERVENTIONS:
Other: 15 subjects with Non Proliferative Diabetic Retinopathy(mild, moderate and severe). 15 subjects with Proliferative Diabetic Retinopathy
  Other Names: NPDR - Non Proliferative Diabetic Retinopathy; PDR -Proliferative Diabetic Retinopathy
  Groups: Diabetic
Other: Healthy Controls 15 age matched control subjects
  Groups: Controls

SUMMARY:
The purpose of this study is to determine if the reparative cells of blood vessels called endothelial progenitor cells(EPC) are defective in people with diabetes.

DETAILED DESCRIPTION:
The purpose of this study is to determine if the reparative cells of blood vessels, called endothelial progenitor cells (EPC's) are defective in people with diabetes. Diabetic retinopathy (DR) is an eye disease related to diabetes. It can cause blurred vision and possible bleeding in the blood vessels in the back of the eye (retina). Damage to the cells of the blood vessels from DR can cause vision loss or blindness. Even with current treatments, the quality of life for people with DR is much reduced.

ELIGIBILITY:
Inclusion Criteria:

* Any man or woman
* Greater than 18 years of age
* Diagnosis of diabetes (applies to the Diabetic Arm only) (N=15 Type 1 and N=15 Type
* The subject must be willing and have the ability to cooperate with the protocol. Children will not be eligible because the investigators need to obtain 150 ml of blood and this is in excess of what can be drawn in children.

Exclusion Criteria:

* Female participants must not be pregnant at the time of the blood draw as evident through a dipstick pregnancy test.
* Have retinal abnormalities other than diabetic retinopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ophthalmology and Primary Care Clinics
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria B Grant, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Diabetic
  15 subjects with Non Proliferative Diabetic Retinopathy(mild, moderate and severe). 15 subjects with Proliferative Diabetic Retinopathy
- Group 2: Healthy Controls
  Healthy Controls 15 age matched control subjects
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 30 | 15
Completed | 30 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 30 | 15 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 15 | 45
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 10 | 30
  Male | 10 | 5 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Increase in Acid Sphingomyelinase (ASM) Expression and Activity in Bone Marrow-derived Endothelial Progenitor Cells (EPCs)
Description: Peripheral blood of 150 cc, about 8-10 tablespoons will be collected from vein in the arm of both diabetic and control subjects.ASM activity was measured on a scale of 0-0.6. 0.6 is worse with units being nM/hr
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: nM/hr
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 30 | 15
nM/hr | 0.2 (0.03) | 0.5 (0.04)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/15
Other Adverse Events (participants affected / at risk) | 0/30 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT03403283/Prot_SAP_000.pdf